CLINICAL TRIAL: NCT05720806
Title: Weight Bearing as Tolerated (WBAT) Following Hip Arthroscopic Labral Repair and Femoroplasty.
Brief Title: Weight Bearing Status Post-hip Arthroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Craig Mauro, Clinical Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY22080053
Record Dates: First submitted 2023-01-10; First posted 2023-02-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hip Impingement Syndrome; Acetabular Labral Tear
MeSH Terms: interventions — Weight-Bearing

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled into either Weight bearing as tolerated group immediately or Flat foot weight bearing group for 2 weeks. Currently, flat foot weight bearing for the first 2 weeks is standard of care.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Physician performing surgical intervention will be blinded from surgery until first follow up. Also, physician performing ultrasound evaluation of hip capsule will remain blinded to weight bearing designation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight bearing as tolerated (WBAT) immediately following surgery. (Experimental): Subjects will be able to self-select weight bearing based on pain and confidence in surgical hip.
  Interventions: Other: Weight Bearing as tolerated (WBAT) immediately following surgery.
- Flat foot weight bearing (FFWB) for 2 weeks after surgery. (Active Comparator): Subjects will be limited to FFWB, approx 20lbs through the surgical hip.
  Interventions: Other: Flat foot weight bearing (FFWB) immediately following surgery

INTERVENTIONS:
Other: Weight Bearing as tolerated (WBAT) immediately following surgery. — Subject will be provided standard of care physical therapy following surgical intervention, except will be able to self-select weight bearing based on pain and confidence.
  Arms: Weight bearing as tolerated (WBAT) immediately following surgery.
Other: Flat foot weight bearing (FFWB) immediately following surgery — Subject will be provided standard of care physcial therapy following surgical intervention except
  Arms: Flat foot weight bearing (FFWB) for 2 weeks after surgery.

SUMMARY:
This study is being proposed to examine weight bearing precautions following hip arthroscopic labral repair, femoroplasty, and capsular closure. Standard post operative protocols limit weight bearing for 2-6 weeks depending on individual surgeons. Cadaveric studies demonstrate that minimal force during weight bearing is distributed through labrum. Therefore, progressing weight bearing earlier in these patients post operatively may help progress faster and improve outcomes. Data collected will include demographic information, radiological data, operative procedures and PRO data.

DETAILED DESCRIPTION:
The study will be conducted at UPMC St. Margaret's Hip Preservation Program. Consented patients who undergo acetabular labral repair and femoroplasty will be included in randomization of weight-bearing status. Two separate protocols will be created to indicate weight bearing status, either WBAT immediately post-op or FFWB immediately post-op, to distribute to rehabilitation staff to ensure compliance. Immediately after the surgical procedure, the surgeon will be blinded and a randomized pamphlet with post-operative instructions with weight bearing education will be given to PACU nursing staff to educate patients and fit crutches.

ELIGIBILITY:
Inclusion Criteria:

* Age>= 12 years
* Diagnoses: femoroacetabular impingement and hip labral tears.
* Surgical procedures performed: Hip arthroscopy with femoroplasty and labral repair.
* Surgery completed at UPMC Children's or UPMC St. Margaret's Hospital
* unilateral and bilateral hip patients

Exclusion Criteria:

* MSK tumor-related FAI or dysplasia
* generalized hypermobility
* revision surgeries

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool 12 (iHot-12) | up to 6 months post-operative
  Scoring ranges from 0-100
  * each question is rated from 0-100 and final score is the mean of all questions answered by subject
  * higher scoring indicating higher quality of life due to hip function
Hip and Groin Outcome Score (HAGOS) | up to 6 months post-operative
  This outcome includes 6 subscales, these are scored independently, and no aggregate scoring is calculated as each section assesses different dimensions separately.
  Subscales (raw scores for each subscale converted to a 0-100 scale with higher score indicating higher level of function):
  * Pain
  * Symptoms
  * Activities of Daily Life
  * Function in Sport and recreation
  * Participation in Physical Activities
  * hip and groin-related quality of life
Hip Outcome Score (HOS) ADL | up to 6 months post-operative
  Outcome assessing function with activities of daily living. Higher score is given for higher level of function and lower score indicating reduced function.
  0-68 aggregate scoring converted to 0-100 scale.
Hip Outcome Score (HOS) Sport | up to 6 months post-operative
  Outcome assessing function/difficulty completing dynamic activities associated with sports participation. Higher score is given for higher level of function and lower score indicating reduced function.
  0-36 aggregate scoring converted to 0-100 scale.
Tampa Scale for Kinesiophobia-11 | up to 6 months post-operative
  Outcome measure assessing fear of pain with movement. Scores range from 11 to 44. Higher scores indicate greater fear of movement

SECONDARY OUTCOMES:
Isometric strength measures hip add, abd, ER, and extension | 6-week, 3 months, and 6-month post-operative
  Strength measures will be taken isometrically at post-operative follow ups.
Diagnostic ultrasound assessment of bilateral anterior hip capsule thickness | 3 months post-operative
  Physician while blinded will perform ultrasound evaluation of the hip capsule to ensure healing.
  Ultrasound will measure the following:
  1.Assess the bilateral hip anterior capsule in all patients, assessing for internal consistency or changes in capsular thickness from side to side. Normal hip capsular thickness has been reported as 7-8 mm, dysplastic hips range 3.2 +/- 0.5 mm, and femoroacetabular impingement subjects 4.7 +/- 0.6 mm.
Diagnostic ultrasound assessment of incision widening | 3 months post-operative
  Physician while blinded will perform ultrasound evaluation of the hip capsule to ensure healing.
  1. Evaluation of capsular incision widening, cyst, attenuation and thinning from established norms. Normal hip capsular thickness has been reported as 7-8 mm, dysplastic hips range 3.2 +/- 0.5 mm, and femoroacetabular impingement subjects 4.7 +/- 0.6 mm
Diagnostic ultrasound for focal echogenic adhesions | 3 months post-operative
  Physician while blinded will perform ultrasound evaluation of the hip capsule to ensure healing.
  1. Evaluate for focal echogenic adhesions or dyskinetic motion between capsule and overlying iliopsoas complex with activation of hip flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Hip Preservation Program, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No